CLINICAL TRIAL: NCT05182476
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of Luvadaxistat in Subjects With Cognitive Impairment Associated With Schizophrenia, Followed by Open-Label Treatment
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Luvadaxistat in Participants With Cognitive Impairment Associated With Schizophrenia
Acronym: ERUDITE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failed to meet the primary endpoint
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1065844-CIAS2023; 2021-003834-34 (EudraCT Number)
Record Dates: First submitted 2021-12-17; First posted 2022-01-10 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive Impairment; Luvadaxistat; NBI-1065844; TAK-831; CIAS; BAC; ERUDITE; Neurocrine
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Drug: Placebo
- Luvadaxistat treatment schedule 1 (Experimental): Luvadaxistat daily
  Interventions: Drug: Luvadaxistat
- Luvadaxistat treatment schedule 2 (Experimental): Luvadaxistat daily
  Interventions: Drug: Luvadaxistat

INTERVENTIONS:
Drug: Placebo — Oral tablets
  Arms: Placebo
Drug: Luvadaxistat — Oral tablets
  Other Names: NBI-1065844; TAK-831
  Arms: Luvadaxistat treatment schedule 1; Luvadaxistat treatment schedule 2

SUMMARY:
Study to evaluate the safety and efficacy of luvadaxistat compared with placebo on improving cognitive performance in participants with schizophrenia.

DETAILED DESCRIPTION:
A Phase 2, randomized, double-blind, parallel, placebo-controlled study with a 6- or 12-month open-label extension. The study is designed to evaluate the efficacy, safety and tolerability, and pharmacokinetics (PK) of treatment with luvadaxistat when administered orally once daily as an adjunctive treatment on improving symptoms of cognitive impairment associated with schizophrenia (CIAS).

ELIGIBILITY:
Key Inclusion Criteria:

Participants must meet all of the following inclusion criteria:

1. Completed written informed consent.
2. Participant must be 18 to 50 years of age (inclusive) and able to comply with all protocol procedures.
3. Diagnosis of schizophrenia as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
4. The initial diagnosis of schizophrenia must be ≥1 year before screening.
5. The participant is currently receiving a stable regimen of psychotropic medications.
6. Participant has stable symptomatology ≥3 months before the screening visit.
7. The participant must have an adult informant.
8. A body weight of at least 45 kilograms (kg) and a body mass index (BMI) of 18.0 to 45.0 kg/meter squared (m^2), inclusive.

Key Exclusion Criteria

Participants will be excluded from the study if they meet any of the following criteria:

1. Pregnant or breastfeeding or plans to become pregnant during the study.
2. Exhibit more than a minimal level of extrapyramidal signs/symptoms.
3. Schizophrenia diagnosis occurred before 12 years of age.
4. Lifetime diagnosis of schizoaffective disorder, bipolar disorder, or obsessive-compulsive disorder.
5. Recent occurrence of panic disorder, depressive episode, or other comorbid psychiatric conditions.
6. Considered by the investigator to be at imminent risk of suicide or injury to self, others, or property, or the participant has attempted suicide within 6 months before screening.
7. Diagnosis of moderate or severe substance use disorder (with the exception of nicotine dependence) within 12 months prior to screening.
8. Positive drug screen for disallowed substances.
9. Any other medical or psychiatric condition or cognitive impairment that may interfere with study conduct or clinical assessments.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Change From Baseline on the Brief Assessment of Cognition in Schizophrenia (BAC) Composite Score | Baseline, Day 98

SECONDARY OUTCOMES:
Change From Baseline on the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Score | Baseline, Day 98
Change From Baseline on the Virtual Reality Functional Capacity Assessment Tool (VRFCAT) | Baseline, Day 98
Change From Baseline on the Clinical Global Impression-Severity Scale (CGI-S) Score | Baseline, Day 98

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (38):
- United States (27):
  - Neurocrine Clinical Site, Phoenix, Arizona
  - Neurocrine Clinical Site, Bentonville, Arkansas
  - Neurocrine Clinical Site, Bryant, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Bellflower, California
  - Neurocrine Clinical Site, Garden Grove, California
  - Neurocrine Clinical Site, Glendale, California
  - Neurocrine Clinical Site, Oceanside, California
  - Neurocrine Clinical Site, Pico Rivera, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, San Rafael, California
  - Neurocrine Clinical Site, Stanford, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Aventura, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Okeechobee, Florida
  - Neurocrine Clinical Site, Pensacola, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Flowood, Mississippi
  - Neurocrine Clinical Site, St Louis, Missouri
  - Neurocrine Clinical Site, Cedarhurst, New York
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, Houston, Texas
- Bulgaria (3):
  - Neurocrine Clinical Site, Pleven
  - Neurocrine Clinical Site, Plovdiv
  - Neurocrine Clinical Site, Sofia
- Czechia (2):
  - Neurocrine Clinical Site, Pilsen
  - Neurocrine Clinical Site, Prague
- Serbia (5):
  - Neurocrine Clinical Site, Belgrade
  - Neurocrine Clinical Site, Gornja Toponica
  - Neurocrine Clinical Site, Kovin
  - Neurocrine Clinical Site, Kragujevac
  - Neurocrine Clinical Site, Niš
- Neurocrine Clinical Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No